CLINICAL TRIAL: NCT02570217
Title: HHHFNC (Heated Humidified High-Flow Nasal Cannula) Versus NCPAP (Nasal Continuous Positive Airway Pressure) in Preterm Infants With Mild to Moderate Respiratory Distress Syndrome (RDS): a Randomized Clinical Trial.
Brief Title: HHHFNC (Heated Humidified High-Flow Nasal Cannula) Versus NCPAP for Respiratory Distress Syndrome of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Dr Anna Lavizzari (Unknown); Dr Francesca Gaia Ciuffini (Unknown)
Responsible Party: Principal Investigator, Mariarosa Colnaghi, MD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHHFNC vs NCPAP 2012; IRCCSMaggioreH (Other: IRCCSMaggioreH)
Record Dates: First submitted 2015-10-03; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Newborn Respiratory Distress Syndrome
Keywords: NCPAP, High Flow Nasal Cannula, pretem infants, NICU
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HHHFNC (Experimental): The patients receive respiratory support by mean of Heated Humidified High Flow Nasal cannula
  Interventions: Device: HHHFNC
- NCPAP (Active Comparator): Patients receive respiratory support by Nasal Continuous Positive Airways Pressure(NCPAP)
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: HHHFNC — infants receive non-invasive respiratory support by mean of HHHFNC
  Other Names: PRECISION FLOW (Vapotherm,Stevensville, USA)
  Arms: HHHFNC
Device: NCPAP — infants receive non-invasive respiratory support by mean of NCPAP
  Other Names: Infant Flow Driver System (EME Ltd, Brighton, Sussex, UK); SiPAP (Viasys Healthcare, Palm Springs, CA)
  Arms: NCPAP

SUMMARY:
Preterm infants ranging from 29+0 to 36+6 weeks+days are randomly assigned to one of the following treatments as non invasive respiratory support if they develop mild to moderate Respiratory Distress Syndrome within 72 hrs from birth: 1) NCPAP set at 4-6 cmH2O or 2) HHHFNC providing a flow 4-6 l/min.

The aim of the study is to assess efficacy and safety of relative "new" form of respiratory support (HHHFNC) versus a more common one (NCPAP).

DETAILED DESCRIPTION:
Preterm infants are eligible to the study if they present mild to moderate Respiratory Distress Syndrome (RDS) defined by the following criteria: need of FiO2 ( Fraction of Inspired Oxygen) ≥0.30 to keep a target SpO2 (Periferal Oxygen Saturation) beetween 88-93% and/or Silverman score ≥5. To confirm the diagnosis a Chest XR is performed as routinarily in the ward before starting the respiratory support.

They are randomly assigned to one of the treatment groups cited in "brief summary" by means of closed envelops. A block randomization is applided with a blok size of 4. The randomization is stratified per groups accoring to gestational age: from 29+0 to 32+6; from 33+0 to 34+6; from 35+0 to 36+6 weeks+days.

Once the treatment is started, for the group NCPAP there is the possibility to switch to the mode "Bi-PAP" if: there are more than 4 episodes of apnoea per hour or more than 2 episodes requiring positive pressure ventilation or if deemed by clinicians for increased work of breathing assesed by the Silverman score.

For all the groups, if the FiO2 requirement is persistently higher than 0.35-0.40 per target SpO2 86-93% and/or dyspnoea defined by Silverman score > 6 after starting the respiratory support, newborns receive Surfactant by "INSURE" technique, involving endotracheal intubation by direct laryngoscopic vision, endotracheal administration of surfactant (Curosurf, Chiesi Pharmaceutics, Parma, Italy) 200 mg/kg and finally extubation.

After the administration of surfactant, if FiO2 requirement is persistently >0.4 to keep SpO2 86-93% or severe apnea episodes are present (apnea episodes > 4/hr or >2/hr requiring positive pressure ventilation) or at the blood gas (capillary or venous) PaCO2>70 mmHg and pH<7.20, newborns are intubated and mechanically ventilated.

For all the newborns enrolled in the study, capillary or venous blood gas is checked every 6-12 hours, a cerebral and cardiac ultrasound screening is performed within 24 hrs. Further controls follow the routine of the ward.

Weaning is started decreasing HHHFNC flow by 1 lpm or nCPAP pressure by 1 cmH2O pressure if infants are presenting FIO2 < 0.30 to target SpO2 and minimal or no signs of respiratory effort. The respiratory support is discontinued for flow ≤ 2 lpm or pressure ≤ 2 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* Inborn
* Parental Consent

Exclusion Criteria:

* No parental consent
* Major congenital malformations
* Severe intra ventricular hemorrage diagnosed early after birth

Ages: 29 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
number of patients needing intubation and mechanical ventilation within 72 hrs from the beginning of the study mode | within 72 hrs from the beginning of the study mode
  The procedure defined as INSURE and described in details in the section "Detailed Study Description" is not considered as a failure for the primary outcome.

SECONDARY OUTCOMES:
overall duration of respiratory assistance | up to 2 years from birth
  respiratory assistance includes both invasive and non invasive respiratory supports
overall duration of oxygen requirement | up to 2 years from birth
  Apart from invasive and non invasive respiratory supports, for this specific outcome are considered also the days of oxygen administration by devices other then ventilators or HHHFNC devices.
overall duration of non invasive respiratory assistance | up to 2 years from birth
  If later during the hospitalisation the newborn receive non invasive ventilation, even if for different reasons from the beginning and/or by mean of a different mode or device, this is registered and computed as "overall non invasive ventilation".
Surfactant treatment | through study completion, an average of 1 year
  the overall number of doses of surfactant are considered
full enteral feeding | through study completion, an average of 1 year
  Number of days required to reach the " full enteral feeding" (defined by a fluids intake about 120 ml/kg/day by enteral administration)
overall duration of hospitalisation | up to 2 years from birth
air-leak syndrome | through study completion, an average of 1 year
Intra ventricular Hemorrage | through study completion, an average of 1 year
Patent Doctus Arterious | through study completion, an average of 1 year
  If a pharmaceutical or surgical treatment is required is considered. Small doctuses closing spontaneously during the first days of life are not included.
Infections | through study completion, an average of 1 year
  Sepsis, pneumonia, cellulites and other infections are considered
Necrotising Enterocolites (NEC) | through study completion, an average of 1 year
Bronchopulmonary Dysplasia | up to 2 years from birth
  Jobe-Bancalari classification criteria are applied.
Retinopathy of Prematurity | through study completion, an average of 1 year
overall mortality | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mariarosa Colnaghi, MD, Study Director — IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
Locations (1):
- NICU, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy, Milan, Italy

REFERENCES:
- [Derived] Lavizzari A, Colnaghi M, Ciuffini F, Veneroni C, Musumeci S, Cortinovis I, Mosca F. Heated, Humidified High-Flow Nasal Cannula vs Nasal Continuous Positive Airway Pressure for Respiratory Distress Syndrome of Prematurity: A Randomized Clinical Noninferiority Trial. JAMA Pediatr. 2016 Aug 8. doi: 10.1001/jamapediatrics.2016.1243. Online ahead of print. PMID 27532363